CLINICAL TRIAL: NCT04460560
Title: A Multi-Center, Open Label, Collaborative Research Study to Treat HRS-AKI Patients With Continuous Terlipressin Infusion
Brief Title: Terlipressin for HRS-AKI in Liver Transplant Candidates (INFUSE)
Acronym: INFUSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 834744
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hepatorenal Syndrome
MeSH Terms: conditions — Hepatorenal Syndrome | interventions — Terlipressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Terlipressin (Other): All prospective patients receive open-label Terlipressin.
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin — For the first dose of terlipressin, each vial will be reconstituted with 5 mL of sterile 0.9% sodium chloride solution and administered intravenously as a bolus injection and given over 1 minute at a dose of 0.5 mg.
  For continuous infusion, the dose of terlipressin is to be dissolved in 0.9% sodium chloride solution and infused with a pump

SUMMARY:
Hepatorenal syndrome-acute kidney injury (HRS-AKI), a potentially reversible renal failure, is a serious, rapidly progressing, often fatal, complication of decompensated cirrhosis. Terlipressin is a synthetic vasopressin analogue that acts as a systemic vasoconstrictor via the vascular vasopressin V1 receptors. In HRS-AKI patients the strong V1 receptor-mediated vasoconstrictor activity of terlipressin, particularly in the splanchnic area, increases effective intravascular volume and mean arterial pressure (MAP), ameliorates renin-angiotensin-aldosterone system and sympathetic nervous system hyperactivity, and improves renal blood flow. The INFUSE trial will evaluate the use of continuous terlipressin infusion in patients on the liver transplant waiting list with HRS-AKI.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent by subject or legally authorized representative.
2. At least 18 years of age.
3. Cirrhosis and ascites.
4. No sustained improvement in renal function (less than 20% decrease in SCr) at least 48 hours after diuretic withdrawal and after plasma volume expansion with albumin (given daily for two days - 48 hours minimum from 1st dose). If SCr improves by ≥ 20 % but plateaus ( ≤ 10 % fluctuation in sCr) and remains above 1.5 mg/dl for ≥another 48 hrs and there are no features of acute tubular necrosis.
5. Increase in SCr by at least ≥ 0.3 mg/dl OR 1.5-2 fold above baseline (AKI stage 1 and above), to a SCr of ≥ 1.5 mg/dl at the time of initiating treatment. Baseline SCr is defined as the most recent, lowest SCr within last 6 months before date of current admission.
6. A.On liver transplant wait list or liver transplant eligible with anticipation of being placed on the liver transplant wait list. B. Patients not on the transplant waitlist or transplant eligible are also eligible for the trial ( maximum 25 subjects) -

Exclusion Criteria:

1. Serum creatinine level greater than 5.0 mg/dL. Subjects with value greater than 5.0 mg/dL may be enrolled with Sponsor prior approval.
2. MELD score ≥ 35
3. Acute on Chronic Liver Failure (ACLF) grade 3 (according to the CLIF Consortium grading system).
4. Uncontrolled sepsis and/or uncontrolled bacterial infection (e.g., persisting bacteremia, persisting ascitic fluid leukocytosis, fever, increasing leukocytosis with vasomotor instability).
5. Shock.
6. Current or recent (within 4 weeks) treatment with or exposure to nephrotoxic agents: eg, aminoglycosides, amphotericin, cyclosporine A, cisplatin, nonsteroidal anti-inflammatory drugs (NSAIDs: e.g., ibuprofen, naproxen, diclofenac), significant exposure to radiographic contrast agents (large doses or multiple injections of iodinated contrast media; e.g., during coronary or abdominal angiogram).
7. Estimated life expectancy of less than 7 days.
8. Advanced Hepatocellular Carcinoma ( HCC) with expected survival of < 6 months
9. Superimposed acute liver injury due to drugs (e.g., acetaminophen), dietary supplements, herbal preparations, viral hepatitis, or toxins (e.g., Amanita toxin with mushroom poisoning carbon tetrachloride), with the exception of acute alcoholic hepatitis.
10. Evidence of obstructive uropathy or parenchymal renal disease. Renal ultrasound or other imaging not required but should be taken if suspicious.
11. Tubular epithelial casts, heme granular casts (range of 1-3 granular casts acceptable), hematuria or microhematuria on urinalysis that is indicative of acute tubular necrosis and/or intrinsic renal disease.
12. Subjects known to be pregnant; all women of child-bearing age and potential must have a negative pregnancy test.
13. Severe cardiovascular disease, including, but not limited to, unstable angina, pulmonary edema, congestive heart failure, or persisting symptomatic peripheral vascular disease, myocardial infarction or stable chronic angina within the past 12 months, or any other cardiovascular disease judged by the investigator to be severe and creates a risk to subject with concurrent terlipressin use.
14. Current or recent (within 4 weeks) renal replacement therapy (RRT) or anticipation of RRT within 3 days on enrollment.
15. Participation in other clinical research involving investigational medicinal products within 30 days of starting study drug that would adversely affect participation in this or the current trial.
16. Transjugular intrahepatic portosystemic shunt (TIPS) within 30 days of starting study drug.
17. For the Prospective Group: All vasopressors must be stopped prior to treatment with terlipressin. Use of vasopressors (e.g., norepinephrine, epinephrine or vasopressin dopamine or other vasopressors) of ≥ 3 consecutive days within the prior 14-day screening period are excluded. Patients receiving a vasopressor other than midodrine within 24 hours of qualifying SCr are excluded, i.e, a 24-h washout is required prior to enrollment.

    Note: Patients receiving midodrine and octreotide may be enrolled. Midodrine and octreotide treatment must be stopped prior to enrollment.
18. Known allergy or sensitivity to terlipressin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - California Pacific Medical Center, San Francisco, California
  - Piedmont Healthcare, Inc, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Prospective Terlipressin Group: Patients to be treated with open label terlipressin by infusion following an initial bolus dose of 0.5mg.
Period: Overall Study
Arm/Group | Prospective Terlipressin Group
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prospective Terlipressin Group
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 59 [28 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 7
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Renal Function (SCr) From Day 1 Thru End of Treatment, Repeated Measure Analysis. SCr Will be Collected Daily, From Day 1 Thru End of Treatment. Baseline SCr Will Also be Entered.
Description: SCr will be collected daily, from Day 1 thru end of treatment. Complete response (CR) defined as ≥30% decrease in SCr with EOT SCr≤1.5, partial response (PR) as ≥30% decrease in SCr with EOT SCr>1.5, and non-response (NR) as <30% decrease in SCr.
Time Frame: 14 days or reversal of HRS-AKI, whichever occur first
Population: descriptive statistics were used only
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Terlipressin: Terlipressin
Arm/Group | Open-label Terlipressin
Number analyzed (Participants) | 50
Participants
  complete response | 32
  partial response | 8
  no response | 10

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Open-Label Terlipressin: All prospective patients receive open-label Terlipressin.
  Terlipressin: For the first dose of terlipressin, each vial will be reconstituted with 5 mL of sterile 0.9% sodium chloride solution and administered intravenously as a bolus injection and given over 1 minute at a dose of 0.5 mg.
  For continuous infusion, the dose of terlipressin is to be dissolved in 0.9% sodium chloride solution and infused with a pump
Arm/Group | Open-Label Terlipressin
All-Cause Mortality (participants affected / at risk) | 14/50
Serious Adverse Events (participants affected / at risk) | 26/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Terlipressin (N=50)
Hypotension (Nervous system disorders) | 3 (3)
AKI (Renal and urinary disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Altered Mental Status (including hepatic encephalopathy) (Nervous system disorders) | 6 (6)
Electrolyte abnormality (Renal and urinary disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multi Organ Failure (General disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Spontaneous Bacterial Peritonitis (Infections and infestations) | 2 (2)
Hepatic hydrothorax (Hepatobiliary disorders) | 1 (1)
Liver failure (Hepatobiliary disorders) | 3 (3)
Peritoneal carcinomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
worsening ascites (Hepatobiliary disorders) | 5 (5)
Decompensated hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04460560/Prot_SAP_000.pdf